CLINICAL TRIAL: NCT07183293
Title: A Multicenter, Randomized, Prospective Study on the Efficacy and Safety of Peginterferon Alfa-2b Combined With Nucleos(t)Ide Analogues in Patients With Compensated HBV-Related Liver Cirrhosis
Brief Title: A Study on Peginterferon Alfa-2b Combined With NAs in Compensated HBV Cirrhosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiamen Humanity Hospital (Other)
Responsible Party: Principal Investigator, Wenqi Huang, Chief physician, Xiamen Humanity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAXM20250731
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: HBV-related Liver Cirrhosis
Keywords: Peginterferon α-2b
MeSH Terms: interventions — nas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: Peginterferon alfa-2b combined with NAs
- Group 2 (Experimental)
  Interventions: Drug: NAs

INTERVENTIONS:
Drug: Peginterferon alfa-2b combined with NAs — Subcutaneous injection therapy,Treatment will continue for 48 weeks, with follow-up assessments conducted every 12 weeks. The dosage will be adjusted based on the patient's disease status.
  Arms: Group 1
Drug: NAs — Treatment will continue for 48 weeks, with follow-up assessments conducted every 12 weeks. The dosage will be adjusted based on the patient's disease status.
  Arms: Group 2

SUMMARY:
This study is a multicenter, randomized, prospective trial designed to evaluate the efficacy and safety of pegylated interferon α-2b (Peg-IFN-α2b) combined with nucleos(t)ide analogues (NAs) versus NAs monotherapy in patients with compensated hepatitis B cirrhosis. A total of 30 patients with compensated HBV-related cirrhosis will be enrolled and randomized in a 2:1 ratio to either Experimental Group 1 (n=20) or Experimental Group 2 (n=10). The treatment regimens consist of Peg-IFN-α2b combined with NAs (ETV/TAF/TMF/TDF) or NAs (ETV/TAF/TMF/TDF) monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of compensated HBV-related liver cirrhosis (Child-Pugh class A or B);
2. The subject is able to understand and comply with the content, requirements, and restrictions of the protocol, is willing and able to complete the study per protocol requirements, fully understands the potential adverse reactions, and voluntarily provides written informed consent prior to study initiation;
3. Aged 18 to 60 years (inclusive), any gender;
4. Female subjects of childbearing potential must have a negative pregnancy test at screening;
5. Subjects (including their partners) must voluntarily use effective non-drug contraception from prior to dosing until six months after discontinuation of the study drug and have no plan to donate sperm or ova; or subjects (including their partners) are of non-childbearing potential (surgically sterilized or postmenopausal).

Exclusion Criteria:

1. Decompensated liver cirrhosis, hepatic failure, or hepatocellular carcinoma; presence of other liver diseases such as fatty liver disease, alcoholic liver disease, drug-induced liver injury, autoimmune liver disease, or Wilson's disease;
2. History of clinically significant diseases of the cardiovascular, hematological and lymphatic, respiratory, urinary, endocrine, immune, psychiatric, or nervous systems (e.g., epilepsy), ophthalmic diseases, or thyroid-related disorders;
3. Pregnancy, lactation, or intention to become pregnant during the study period;
4. Known or suspected allergy to the investigational product(s) or any of its excipients;
5. Participation in any other interventional clinical trial within 3 months prior to screening or planning to participate in another clinical trial during the study;
6. Any other condition considered by the investigator to be inappropriate for participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Change in liver histological score from baseline | 24 weeks after the end of treatment

SECONDARY OUTCOMES:
Incidence of hepatocellular carcinoma (HCC) | Week 48
Incidence of hepatic decompensation events | Week 48
Change in liver stiffness measurement (LSM) from baseline | Week 48,24 weeks after the end of treatment
  Evaluation is performed using liver imaging data such as liver MRI and histopathological data.
Change in AST-to-Platelet Ratio Index (APRI) from baseline | Week 48,24 weeks after the end of treatment
Change in Fibrosis-4 Index (FIB-4) from baseline | Week 48,24 weeks after the end of treatment
HBsAg loss rate | Week 48,24 weeks after the end of treatment
Seroconversion rate | Week 48,24 weeks after the end of treatment
HBeAg loss rate | Week 48,24 weeks after the end of treatment
HBV DNA undetectability rate | Week 48,24 weeks after the end of treatment
HBV RNA undetectability rate | Week 48,24 weeks after the end of treatment
HBV RNA decline rate | Week 48,24 weeks after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wenqi Huang, Principal Investigator — Xiamen Humanity Hospital
Locations (2):
- China (2):
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen

IPD SHARING:
Plan to Share IPD: No